CLINICAL TRIAL: NCT01903083
Title: Phase I Trial of Chemoimmunotherapy and Hypofractionated Radiation Therapy for Borderline Resectable and Locally Advanced Pancreatic Adenocarcinoma.
Brief Title: Chemoimmunotherapy and Radiation in Pancreatic Cancer
Acronym: CRIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-026A
Record Dates: First submitted 2013-07-02; First posted 2013-07-19 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Locally Advanced Malignant Neoplasm
Keywords: Pancreas; Pancreatic cancer; Immunotherapy; Chemotherapy; Radiation; Surgery; Pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Tadalafil; Gemcitabine; Radiation; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunochemoradiotherapy (Experimental): Immunotherapy with oral tadalafil daily; three doses of chemotherapy with IV Gemcitabine in 21-day cycles for up to 4 cycles; three fractions of external beam radiation to the pancreas and and regional lymph nodes; pancreaticoduodenectomy (surgical resection) for eligible patients.
  Interventions: Drug: Tadalafil; Drug: Gemcitabine; Radiation: Radiation; Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Drug: Tadalafil — One 2.5 mg tablet is self-administered orally by the study participant on a once daily basis.
  Other Names: Cialis
Drug: Gemcitabine — Three doses of gemcitabine (1000 mg / m^2)are given over a 21-day cycle. Patients may receive up to 4 cycles.
  Other Names: Gemzar
Radiation: Radiation — Patients will receive 3 doses of radiation (8-10 Gy per fraction).
Procedure: Pancreaticoduodenectomy — Surgical resection.

SUMMARY:
The goal of this study is to evaluate the safety of combination treatment that includes chemotherapy, radiation therapy, and immunotherapy in patients with pancreatic cancer.

DETAILED DESCRIPTION:
This study is for borderline resectable and advanced pancreatic cancer patients. Patients will receive chemotherapy with gemcitabine and immunotherapy with daily tadalafil during the first 21 days of treatment. On study day 22, patients will receive the first of three planned doses of radiation therapy and continue daily tadalafil. Patients are then evaluated to determine if they are candidates for pancreaticoduodenectomy. Patients who are not candidates will continue daily tadalafil and receive gemcitabine chemotherapy. Patients who have surgery will resume daily tadalafil and gemcitabine chemotherapy following recovery from surgery. Patients will receive up to four cycles of gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic adenocarcinoma
* Locally advanced unresectable disease, or borderline resectable disease
* ECOG (Eastern Cooperative Oncology Group)Performance Status 0 or 1
* Ability to provide consent and comply with study protocol
* Women of child-bearing potential must have a negative pregnancy test and avoid pregnancy during the study

Exclusion Criteria:

* Age < 18
* History of other malignancy in previous 2 years except carcinoma in situ of the cervix or bladder, or non-melanoma skin cancer
* Previous chemotherapy or radiation therapy for pancreatic cancer or previous radiation to the target field
* Clinically active autoimmune disease or active infection
* History of heart attack within 90 days or stroke within 6 months, hypertension requiring change in blood pressure medications in the last 4 weeks, hypotension, uncontrolled arrhythmias, heart failure (NYHA >= Class 2 in last 6 months), unstable angina, or angina during sexual activity
* Use of nitrates or nitroglycerin
* History of hereditary degenerative retinal disorders including retinitis pigmentosa
* Chronic systemic corticosteroid use at supra-physiologic doses
* Use of recreational drugs called 'poppers' like amyl nitrite and butyl nitrite
* Blood test results (neutrophils < 1000 /uL (microliter); hemoglobin < 9 gm /dL; platelet count < 1000 cells / uL; significant coagulopathy; significant liver or renal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety | 135 Days
  Patients will return be seen in the clinic 8 times over the first 50 days for an evaluation of adverse events and toxicities before being evaluated for surgery. Patients who are not candidates for surgery will be seen in clinic 10 more times over the next 85 days for safety evaluations, and patients who have surgery will be seen 10 times over the 85 days following recovery from surgery for safety evaluations.

SECONDARY OUTCOMES:
Immune Infiltration in pancreaticoduodenectomy tissue | 50 Days
  For surgery patients, formalin fixed and paraffin-embedded tumor tissue obtained during surgery will be sectioned and immunohistology performed to determine the tumor inflammatory micro-environment and the degree of macrophage and T cell inflammation.
Quantification of T cells in peripheral blood pre- and post-treatment | 135 Days
  Patients will provide a pre-treatment blood sample and 4 blood samples over 135 days to evaluate the influence of the study treatment on immune parameters. For patients who have surgery, the time period will be longer depending on their recovery time. Post-treatment long term follow up will occur every 12 weeks (+/- 2 weeks) beyond post-recovery date (PRD) 85 for 6 visits. Blood will be collected for immune monitoring at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Crocenzi, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crocenzi T, Cottam B, Newell P, Wolf RF, Hansen PD, Hammill C, Solhjem MC, To YY, Greathouse A, Tormoen G, Jutric Z, Young K, Bahjat KS, Gough MJ, Crittenden MR. A hypofractionated radiation regimen avoids the lymphopenia associated with neoadjuvant chemoradiation therapy of borderline resectable and locally advanced pancreatic adenocarcinoma. J Immunother Cancer. 2016 Aug 16;4:45. doi: 10.1186/s40425-016-0149-6. eCollection 2016. PMID 27532020